CLINICAL TRIAL: NCT00642096
Title: A Phase III, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Factorial Study of Metoprolol Succinate Extended Release Tablets (TOPROL-XL) Hydrochlorothiazide and Their Combination in Patients With Essential Hypertension.
Brief Title: Factorial Study of Metoprolol Succinate TOPROL-XL (324A)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D4026C00001
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: High Blood Pressure (Hypertension).
Keywords: High blood pressure; hypertension; (TOPROL-XL); metoprolol succinate; hydrochlorothiazide
MeSH Terms: conditions — Hypertension | interventions — Metoprolol; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Metoprolol Succinate + Hydrochlorothiazide
  Interventions: Drug: Metoprolol Succinate; Drug: Hydrochlorothiazide
- 2 (Active Comparator): Metoprolol Succinate
  Interventions: Drug: Metoprolol Succinate
- 3 (Active Comparator): Hydrochlorothiazide
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Metoprolol Succinate
  Other Names: TOPROL-XL
  Arms: 1; 2
Drug: Hydrochlorothiazide
  Arms: 1; 3

SUMMARY:
The purpose of this research study is to determine if treatment with the combination of metoprolol succinate and hydrochlorothiazide is more effective at lowering blood pressure than treatment with either of the two drugs alone. The study will also determine which combined doses of metoprolol succinate and hydrochlorothiazide are most effective at lowering blood pressure (without unacceptable side effects), and whether it is possible to combine both drugs in a single tablet to simplify blood pressure treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diastolic blood pressure between 95 and 114 mm at screening and start of treatment

Exclusion Criteria:

* Significant conditions which in the opinion of the investigator place the subject at undue risk, eg Renal impairment, hepatitis
* Known secondary causes of hypertension, eg, Cushing's syndrome, renal artery stenosis, pheochromocytoma, hyperaldosteronism
* Systolic blood pressure greater or equal to 180 mm Hg at start of trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1900 (Estimated)
Dates: Start 2003-06; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Change in trough sitting diastolic blood pressure | 3 readings determined at 8 weeks after treatment

SECONDARY OUTCOMES:
change in trough Sitting Systolic Blood pressure | 3 readings determined at 8 weeks after treatment
change in trough Standing Systolic Blood Pressure | 6 readings determined at 8 weeks after treatment
change in trough standing diastolic blood pressure | 6 readings determined at 8 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Vasilios Papademetriou, Principal Investigator — Georgetown University